CLINICAL TRIAL: NCT00530179
Title: FDG-PET-Stratified R-DICEP and R-BEAM/ASCT For Diffuse Large B-Cell Lymphoma
Acronym: PET-Chop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Douglas Stewart, Dr. Douglas Stewart - Principal Investigator, AHS Cancer Control Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0307003
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma; Positron Emission Tomography; CHOP Chemotherapy protocol; Stem Cell Transplantation; Fluorodeoxyglucose F18
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Standard R-CHOP chemotherapy every 21 days X 2 Cycles followed by PET/CT scan. If scan is determined negative for disease intensity patient receives 4 more cycles R-CHOP (total 6 cycles R-CHOP)
  Assigned interventions: Drug: R-CHOP (Rituximab, Cyclophosphamide, Etoposide, Cisplatin, Mesna, G-CSF 6 - 21 DAY Cycles of R-CHOP
  Interventions: Drug: R-CHOP
- Arm B (Active Comparator): Standard R-CHOP chemotherapy every 21 days X 2 Cycles followed by PET/CT scan. If scan is determined positive for disease intensity the patient receives one cycle or R-DICEP/R-BEAM the autologous blood stem cell transplantation.
  Assigned Interventions: Procedure/Surgery: Autologous Blood Stem Transplantation 2 CYCLES OF R-CHOP + R-DICEP/R-BEAM FOLLOWED BY AUTOLOGOUS BLOOD STEM CELL TRANSPLANTATION
  Interventions: Procedure: Autologous Blood Stem Transplantation

INTERVENTIONS:
Procedure: Autologous Blood Stem Transplantation — 2 CYCLES OF R-CHOP + R-DICEP/R-BEAM FOLLOWED BY AUTOLOGOUS BLOOD STEM CELL TRANSPLANTATION
  Arms: Arm B
Drug: R-CHOP — 6 - 21 DAY Cycles of R-CHOP
  Arms: Arm A

SUMMARY:
The purpose of this study is to evaluate:

1. whether an imaging test called a PET (Positron emission tomography) scan performed after two cycles of standard chemotherapy is able to identify patients who have a high cure rate after completing standard chemotherapy alone; and
2. whether high dose chemotherapy (HDCT) and autologous stem cell transplantation (ASCT) when used in combination with an antibody called Rituximab results in high cure rates for those patients predicted to do poorly with standard chemotherapy by the PET scan.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Although the addition of Rituximab anti-CD20 monoclonal antibody therapy to standard CHOP chemotherapy (R-CHOP) results in a 15-20% increase in absolute EFS rate over CHOP alone for DLBCL patients, it is likely that 40-50% of patients with poor prognosis DLBCL will not be cured by R-CHOP. High dose chemotherapy (HDCT) and autologous stem cell transplantation (ASCT) has been shown to salvage a substantial proportion of patients with relapsed DLBCL. A meta-analysis of randomized controlled trials comparing standard-dose chemotherapy (SDCT) alone to SDCT followed by HDCT/ASCT as initial treatment for poor prognosis DLBCL demonstrated a significant benefit for HDCT over SDCT in terms of EFS and OS. A single centre prospective phase II study was conducted in Calgary to assess feasibility, toxicity, and efficacy of two cycles of HDCT following just one cycle of CHOP induction therapy for patients under 65 years of age who were diagnosed with aggressive histology lymphoma and 2-3 Age Adjusted International Prognostic Index (AAIPI) risk factors. The study was conducted prior to the widespread use of Rituximab plus CHOP (R-CHOP). The treatment protocol involved one cycle of standard dose CHOP followed by one cycle of dose-intensive cyclophosphamide 5.25 g/m2, etoposide 1.05 g/m2, cisplatin 105 mg/m2 (DICEP), then autologous blood stem cell collection, followed by one cycle of high dose BCNU 300 mg/m2, etoposide 800 mg/m2, Ara-C 1600 mg/m2, melphalan 140 mg/m2 (BEAM) and autologous stem cell transplantation (ASCT) and radiotherapy to prior bulk. With a median follow up of 49 months, 4 year event free (EFS) and overall survival (OS) rates for the 55 patients accrued to the study were 72% (95% CI=60-84%) and 79% (95% CI=69-90%), respectively.

The two major advances in lymphoma management that have occurred since the design of our CHOP-DICEP-BEAM/ASCT phase II study are the addition of Rituximab anti-CD20 monoclonal antibody therapy to chemotherapy (as described above), and the use of FDG-PET functional imaging/response assessment. Several studies have reported the strong correlation of early response assessment using FDG-PET with PFS and OS following standard chemotherapy for aggressive NHL. In one of the largest, best designed studies, PET-negativity following 2 cycles of RCHOP was associated with higher 2-year estimates of EFS (82% vs 43% , p < .001) and OS (90% vs 61%, p = .006). The incorporation of Rituximab and PET-guided HDCT/ASCT into our intensive chemotherapy protocol may lead to further improvements in EFS while decreasing the overall need for HDCT/ASCT by targeting those patients destined to fail R-CHOP by early PET-based response assessment.

STUDY OBJECTIVES:

1. To determine if negative FDG-PET imaging following 2 cycles of R-CHOP chemotherapy is able to identify a group of patients with excellent prognosis (80% 3-year EFS) following standard 6 cycles of R-CHOP chemotherapy alone.
2. To determine if a group of patients with positive FDG-PET imaging following 2 cycles of R-CHOP chemotherapy are able to achieve excellent outcome (80% 3-year EFS) following intensive chemotherapy with R-DICEP and R-BEAM/ASCT.
3. To determine if PET-guided R-DICEP and R-BEAM/ASCT is feasible and associated with acceptable toxicity rates in a multi-centre study.

STUDY DESIGN:

INCLUSION CRITERIA:

1. Give written informed consent
2. Age 18-65 years
3. Histological diagnosis of Diffuse Large B-cell Lymphoma including:

   1. Diffuse Large B-cell
   2. Immunoblastic B-cell
   3. Primary Mediastinal Diffuse Large B-cell
   4. T-cell Rich, Diffuse Large B-cell
   5. Anaplastic Large B-Cell
   6. Diffuse Large B-cell with areas of follicular lymphoma in same biopsy
4. No central nervous system involvement by lymphoma
5. No more than 1 prior cycle of R-CHOP chemotherapy
6. At least 1 adverse International Prognostic Index factor at diagnosis:

   a. Age > 60 years b. ECOG performance status 2-4 c. Elevated serum LDH level d. More than 1 extranodal site involved by lymphoma e. Stage 3 or 4
7. Adequate organ function:

   1. Cardiac: LVEF >45%
   2. Pulmonary: FVC, FEV1 and DLCO >50% predicted
   3. Renal: creatinine <120µmol/L unless caused by ureteric obstruction from lymphoma
   4. Liver: ALT, AlkP, Bilirubin <3 x upper limit of normal unless caused by biliary tract obstruction from lymphoma

      EXCLUSION CRITERIA:

      1. Histological diagnosis other than Diffuse Large B-cell Lymphoma 2. Pregnant or lactating females 3. Concurrent use of other anti-cancer therapies 4. Other serious co-morbid illness that would compromise study participation. 5. Prior malignancy unless non-melanoma skin cancer, carcinoma in-situ of the cervix (CIN) or breast, or malignancy treated more than 5 years previously with no evidence of recurrent disease since initial treatment.

      6. More than 1 prior cycle of Rituximab, cyclophosphamide, or doxorubicin. 7. Prior HDCT/ASCT or prior radiotherapy.

      STUDY ENDPOINTS

      Primary:

      • 3 year EFS for patients receiving 6 cycles R-CHOP (PET-negative response) and for patients receiving RCHOP x2 followed by R-DICEP then R-BEAM/ASCT (PET-positive response)

      Secondary:

      • Complete and Partial Response Rates

      • PET/CT response rates following RCHOP x 2 cycles

      • Overall Survival
      * Safety (type, frequency, severity, and relationship of adverse events to study treatment)

      STUDY DURATION: Three years TOTAL SAMPLE SIZE: 70-80 patients

      DOSING REGIMEN(S):

<!-- -->

1. Induction: Standard R-CHOP chemotherapy q21days x 2 cycles

   R-CHOP x 2 cycles q21days:

   Rituximab 375mg/ m2 IV day 1 Cyclophosphamide 750mg/ m2 IV day 1 Adriamycin 50mg/ m2 IV day 1 Vincristine 1.4mg/ m2 (max 2mg) IV day 1 Prednisone 100mg po days 1-5
2. FDG-PET/CT imaging between days 10-15 following R-CHOP cycle #2.

Sites of disease will be scored for intensity based on the following scale:

1. Absent
2. Minimal (low grade but greater than in regional lymph nodes of similar size or surrounding interstitial tissues)
3. Low (readily visible but less than liver)
4. Medium (comparable to liver)
5. High (greater than liver)

   Interim post therapy scans will be considered as negative (showing a favorable response) if no more than one site shows an intensity score of greater than 3.

   The treatment protocol will be dictated by the result of the interim FDG-PET/CT scan following 2 cycles of R-CHOP chemotherapy as follows:
   1. If FDG-PET scan negative: 4 more cycles R-CHOP (total 6 cycles R-CHOP)
   2. If FDG-PET scan positive: one cycle of R-DICEP then within 5-8 weeks administer R-BEAM and autologous blood stem cell transplantation as outlined below:

      3) For PET-positive patients ONLY:

   R-DICEP CHEMOTHERAPY (begin 3-5 weeks following day 1 CHOP #2).

   ½NS+20meq KCL/L IV at 150ml/h start 19:00h day 1 then decrease to 75ml/h at 08:00am day 2, continue to day 5 Rituximab 375mg/m2 IV day 1 and 8 (day 1 on a Wednesday) Cyclophosphamide 1.75 g/ m2 d2,3,4 in 500ml D5W over 2 hrs Etoposide 350 mg/ m2 d2,3,4 in 1 L over 2 hrs daily Cisplatin 35 mg/m2 d2,3,4 in 500ml N/S +25g mannitol over 2 hrs Mesna 1.75g/m2 d2,3,4 by continuous infusion over 24 hrs G-CSF 300 (<70kg), 480 (70-100kg), or 600mcg/d (>100kg) SC from day 15 until apheresis completed

   AUTOLOGOUS BLOOD STEM CELL COLLECTION:

   Apheresis approximately day 20-22 of R-DICEP, after ANC>5 x 109/L, platelets increasing >50 x109/L , and peripheral blood CD34 count >20 x106/L (if measurement available). Apheresis to proceed according to standards set at each study centre until at least 3x106CD34+ cells/kg have been collected (>5x106 CD34+ cells/kg preferred).

   R-BEAM + Autologous Stem Cell Transplantation (5-8weeks post-d1 R-DICEP)

   Day - 6 Rituximab 375mg/m2 IV BCNU 300mg/m2 IV Day -5 to -2 Etoposide 100mg/m2 IV q12h x 8 doses Ara-C 200mg/m2 IV q12h x 8 doses Day -1 Melphalan 140mg/m2 IV Day 0 Stem Cell Infusion Day 14 Rituximab 375mg/m2 IV

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of Diffuse Large B-Cell Lymphoma
* Adverse Prognosis = Stage 3 or 4 and elevated LDH
* No more than one prior cycle of R-CHOP chemotherapy
* Adequate cardiac function
* No central nervous system involvement by lymphoma

Exclusion Criteria:

* Histological diagnosis other than Diffuse Large B-cell Lymphoma
* Pregnant or lactating females
* Use of other anti-cancer therapies
* Other serious illness that would compromise study participation
* Prior malignancy
* Prior stem cell transplant or radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-07; Primary Completion 2014-02 (Actual); Study Completion 2015-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Stewart, M.D., Principal Investigator — AHS Cancer Control Alberta
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Ottawa General Hospital, Ottawa, Ontario
  - Saskatchewan Cancer Agency, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No